CLINICAL TRIAL: NCT01983410
Title: A Registry for BRCA Mutation Carriers With Pancreatic Ductal Adenocarcinoma
Status: Active, not recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Abramson Cancer Center at Penn Medicine (Other); Shaare Zedek Medical Center (Other); Sheba Medical Center (Other Government); Dana-Farber Cancer Institute (Other); Johns Hopkins University (Other)
Responsible Party: Sponsor
Other Study IDs: 13-217
Record Dates: First submitted 2013-11-04; First posted 2013-11-14 (Estimated); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Pancreatic Ductal Adenocarcinoma
Keywords: BRCA Mutation Carriers; PDAC carriers; BRCAmut carriers; Registry; 13-217

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — Blood specimens tumor tissue samples will be requested

GROUPS / COHORTS (5):
- BRCAmut carrier relatives of a BRCAmut PDAC patient: Who themselves have no known prior or active personal history of non-PDAC malignancy (e.g. breast , ovarian cancer or prostate cancer)
  Interventions: Behavioral: The risk assessment questionnaire; Other: Blood specimens
- BRCAmut carrier relatives of a BRCA mutation PDAC: Patient who themselves have a known prior or active breast, ovarian cancer or prostate cancer
  Interventions: Behavioral: The risk assessment questionnaire; Other: Blood specimens
- BRCAmut carriers: who are not related to a BRCAmut PDAC patient
  Interventions: Behavioral: The risk assessment questionnaire; Other: Blood specimens; Other: tumor tissue samples will be requested
- AJ PDAC patients: who are proven non-BRCAmut carriers.
  Interventions: Behavioral: The risk assessment questionnaire; Other: Blood specimens; Other: tumor tissue samples will be requested
- AJ first or second degree relatives of an AJ PDAC patient from a multiplex family: A family with at least two first or second degree relatives w ho have had PDAC.
  Interventions: Behavioral: The risk assessment questionnaire; Other: Blood specimens; Other: tumor tissue samples will be requested

INTERVENTIONS:
Behavioral: The risk assessment questionnaire
Other: Blood specimens
Other: tumor tissue samples will be requested
  Groups: AJ PDAC patients; AJ first or second degree relatives of an AJ PDAC patient from a multiplex family; BRCAmut carriers

SUMMARY:
The purpose of this study is to better understand why pancreatic cancer develops in some people who are known carriers of the gene mutation (an abnormality) called BRCA, or its close relative PALB2. The investigators hope to do this by establishing a BRCA/PALB2 mutation carriers Pancreatic Ductal Adenocarcinoma (the common form of pancreatic cancer) Registry. A registry is a database of information.

ELIGIBILITY:
Inclusion Criteria:

* BRCA mutation carrier is defined as a person with any mutation of the BRCA gene, including BRCA1, or BRCA2. PALB2mut patients are also eligible.
* Relative of a BRCA PDAC patient is defined as a first-degree relative, which includes, parents, siblings or children.

BRCAmut PDAC Group: Study Group A: Ashkenazi Jewish descent

* Known BRCA mutation carrier.
* Ashkenazi Jewish Descent (at least one parent of Ashkenazi Jewish origin).
* Histologic proof of primary pancreatic ductal adenocarcinoma.
* May have either potentially curable (resectable) primary PDAC, localized but unresectable primary PDAC, or metastatic (stage IV) PDAC.
* Prior personal history of other malignancy; either prior or currently active, including breast , ovarian or prostate cancer is allowed.
* Both previously treated and previously untreated patients are eligible. Previous treatment may include surgical resection, regional radiation therapy, or systemic therapy. Patient may be receiving active therapy.
* Willing to provide blood specimens for correlative studies.
* Willing to provide permission to obtain banked tumor tissue for analysis (previous biopsies or surgical material). New tumor biopsies are not required for entrance into the Registry.

BRCAmut PDAC Group: Study Group B: non-Ashkenazi Jewish descent

* Know n BRCA mutation carrier.
* Histologic proof of primary pancreatic ductal adenocarcinoma.
* May have either potentially curable (resectable) primary PDAC, localized but unresectable primary PDAC, or metastatic (stage IV) PDAC.
* Prior personal history of other malignancy; either prior or currently active, including breast, ovarian, or prostate cancer is allowed.
* Both previously treated and previously untreated patients are eligible. Previous treatment may include surgical resection, regional radiation therapy, or systemic therapy. Patient may be receiving active therapy.
* Willing to provide blood specimens for correlative studies.
* Willing to provide permission to obtain banked tumor tissue for analysis (previous biopsies or surgical material). New tumor biopsies are not required for entrance into the Registry.

BRCA mutation carrier, relative of a BRCA PDAC patients, without PDAC or other BRCAmut related malignancy: (Control Cohort 1A): Ashkenazi Jewish descent

* Known BRCA mutation carrier.
* Ashkenazi Jewish Descent (at least one parent of Ashkenazi Jewish origin).
* No current or prior history of PDAC.
* Relative of a BRCAmut PDAC patient; no prior or active personal history of breast, ovarian, or prostate cancer
* Willing to provide blood specimens for correlative studies.

BRCA mutation carrier, relative of a BRCA PDAC patients, without PDAC or other BRCAmut related malignancy: (Control Cohort 1B): non-Ashkenazi Jewish descent

* Know n BRCA mutation carrier.
* No current or prior history of PDAC.
* First or second degree relative of a BRCAmut PDAC patient; no prior or active personal history of breast, ovarian, or prostate cancer.
* Willing to provide blood specimens for correlative studies.

BRCAmut Carrier relative of a BRCAmut PDAC patient who themselves have prior or active BRCAmut related malignancy (Control Cohort 2A):Ashkenazi Jewish descent

* Known BRCA mutation carrier.
* Ashkenazi Jewish Descent (at least one parent of Ashkenazi Jewish origin).
* No current or prior history of PDAC.
* Relative of a BRCAmut PDAC patient.
* Prior or active personal history of any BRCA-related cancer.
* Willing to provide blood specimens for correlative studies.

BRCAmut Carrier relative of a BRCAmut PDAC patient who themselves have prior or active BRCAmut related malignancy (Control Cohort 2B): non-Ashkenazi Jewish descent

* Know n BRCA mutation carrier.
* No current or prior history of PDAC.
* First or second degree relative of a BRCAmut PDAC patient.
* Prior or active personal history of any BRCA-related cancer.
* Willing to provide blood specimens for correlative studies.

BRCAmut carrier who is not related to a BRCAmut PDAC patient: (Control cohort 3A) Ashkenazi Jewish descent

* Known BRCAmut carrier.
* Ashkenazi Jewish decent (at least one parent of Ashkenazi Jewish origin).
* No current or prior personal history of PDAC.
* Prior personal history of other malignancy including breast, ovarian or prostate cancer is allowed.
* Willing to provide blood specimens for correlative studies.

BRCAmut carrier who is not related to a BRCAmut PDAC patient: (Control cohort 3B) non-Ashkenazi Jewish descent

* Know n BRCAmut carrier.
* No current or prior personal history of PDAC.
* Prior personal history of other malignancy including breast, ovarian, or prostate cancer is allowed.
* Willing to provide blood specimens for correlative studies.

Non-BRCAmut carriers with histologically proven PDAC: (Control cohort 4) Tested for and negative for the BRCA founder mutations.

* Ashkenazi Jewish Descent (at least one parent of Ashkenazi Jewish origin).
* Not related to known BRCAmut carrier.
* Histologic proof of primary pancreatic ductal adenocarcinoma. May have either potentially curable (resectable) primary PDAC, localized but unresectable primary PDAC, or metastatic (stage IV) PDAC.
* Both previously treated and previously untreated patients are eligible. Previous treatment may include surgical resection, regional radiation therapy, or systemic therapy. Patient may be receiving active therapy.
* Willing to provide blood specimens for correlative studies.
* Willing to provide permission to obtain banked tumor tissue for analysis (previous biopsies or surgical material). New tumor biopsies are not required for entrance into the Registry

Exclusion Criteria:

* Individuals will be excluded from the Registry if they:
* Are unable to sign informed consent for medical or other reasons. Do not speak English (MSK and UPenn) or do not speak English or Hebrew (BCGC Sites).
* Are under 21 years of age.
* Not willing to provide blood samples for correlative studies.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: BRCA mutation carriers with PDAC will be identified by the PIs, co-investigators and by the research staff at all participating sites.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2013-11-04 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
prospective Registry | 3 years
  Establishment of a BRCA mutation carriers PDAC Registry with appropriate control groups, and collection and storage of biological material for future studies.

CONTACTS AND LOCATIONS:
Overall Officials: David Kelsen, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (13):
- United States (10):
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Cold Springs Harbor Laboratory (Specimen Analysis), Cold Spring Harbor, New York
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Weill Cornell Medical College (Specimen Analysis), New York, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York
  - Abramson Cancer Center at University of Pennsylvania Medical Center, Philadelphia, Pennsylvania
- Israel (3):
  - Shaare Zedek Medical Center, Jerusalem
  - Weizmann Institute of Science (Specimen Analysis), Rehovot
  - Sheba Medical Center, Tel Litwinsky

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/